

#### **PARTICIPANT INFORMATION SHEET**

Please read the following information carefully. Do not hesitate to discuss any questions you may have with your doctor.

### **Study Title**

Evaluation of The Kotak as a School-Based Smoking Prevention and Intervention Programme in Malaysian Public School

#### Introduction

Smoking is a public health concern. It is associated with many diseases including oral diseases. Recognising the importance to prevent smoking, the Oral Health Division, Ministry of Health has implemented a school-based smoking prevention and quit smoking programme among primary and secondary schoolchildren through its school dental service. This programme is known as KOTAK. The aims of the KOTAK programme is to provide brief and advance intervention to stop smoking to those schoolchildren who are smokers. It is important to evaluate the effectiveness of this programme as to provide evidence of the worth of implementing such programme in reducing the prevalence of smoking among schoolchildren.

### What is the purpose of this study?

The purpose of this study is to evaluate the impacts the KOTAK programme has on smoking cessation success among adolescents.

#### What are the procedures to be followed?

Each participant is required to answer a set of questionnaires related to their exposure to cigarettes and to undergo a clinical oral examination.

Each participant is also required to exhale their breath in a device that record the carbon monoxide level. In addition, a sample of saliva of no less than 2ml is required from each participant.

### Who should not enter the study?

Secondary schoolchildren who is not medically and physically fit to participate in this study. This include those who did not have parental consent.

### What will be the benefits of the study?

- (a) To participant?
  - There are no direct benefits for the participants enrolling into this research. However, your participation will indeed benefit the society at large.
- (b) To the investigator?

Your response will help the investigators to analyse and provide an evidence to the respective authorities to plan a comprehensive programme in the future pertaining to the implementation of the KOTAK programme.

### What are the possible drawbacks? / risks / complications / adverse effects that may happen?

Your participation is entirely voluntary. There are no drawbacks. You can withdraw your participation at any time and the refusal will not affect your schooling.

### Can I refuse to take part in the study?

Your participation is totally voluntary. You need not have to explain why you prefer not to take part in the study.

Who shall I contact if I have additional questions/complications during the course of the study?

Main and other investigators (all listed in the application form):

(1) Investigator's Name:



### CONSENT BY PARTICIPANT FOR RESEARCH FACULTY OF DENTISTRY, UM, K.L.

| I, | rd No |
|---|---|
| of | |
| Title of Study: | |
| Evaluation of The Kotak as a School-Based Smoking Prevention and Intervention Programme in Malaysian Public School | |
| The nature and purpose of the research has been explained to me by XXX, Researcher and interpreted (when necessary) by | |
| I understand that I can withdraw from this research at any time without assigning my reason whatsoever. | |
| Signature(Participant) | Date |
| IN THE PRESENCE OF | |
| Name, | |
| I/C No, | Position |
| Signature(Witness for signature of participant) | Date |
| I confirm that I have explained to the participant the nature and purpose of the above-mentioned research. | |
| Signature (Attending doctor) | Date |



### CONSENT BY PARTICIPANT'S PARENT/GUARDIAN FOR RESEARCH FACULTY OF DENTISTRY, UM, K.L.

| I, of *(Name of participant's parent/guardian) |
|---|
| hereby agree |
| (Address) |
| to allow my daughter/son named to take part in the (Name of participant) |
| research specified below: |
| Title of Study: |
| Evaluation of The Kotak as a School-Based Smoking Prevention and Intervention Programme in Malaysian Public School |
| After knowing and understanding all the possible advantages and disadvantages of this research, I voluntarily consent of my own child to participate. |
| I understand that my child can withdraw from this research at any time. |
| Signature Date |
| *(Participant's parent/ guardian) |
| (rantospanico parone gadraran) |
| IN THE PRESENCE OF |

